CLINICAL TRIAL: NCT01470521
Title: Worms for Immune Regulation of Multiple Sclerosis (WIRMS)
Brief Title: Worms for Immune Regulation of Multiple Sclerosis
Acronym: WIRMS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08126
Record Dates: First submitted 2011-11-09; First posted 2011-11-11 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Multiple sclerosis; Hookworm larvae; Necator americanus; Treg cells
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — ASP-1 protein, Necator americanus; Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hookworm larvae (Necator americanus) (Experimental): Participants will receive 25 live hookworm larvae
  Interventions: Biological: Hookworm larvae
- Placebo (Placebo Comparator): Participant will receive pharmacopoeial grade water
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Hookworm larvae — Hookworm larvae solution is pipetted onto a plaster dressing which is then placed on the upper forearm for 24 hours. This is administered only once.
  Other Names: Necator americanus
  Arms: Hookworm larvae (Necator americanus)
Biological: Placebo — Pharmacopoeial grade water is pipetted onto a plaster dressing which is then placed on the upper forearm for 24 hours. This is administered only once.
  Other Names: Water
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether people with MS who are exposed to a small number of hookworms will have less inflammation and less MS disease activity.

DETAILED DESCRIPTION:
There is evidence that certain parasitic infections may protect against autoimmune or inflammatory diseases, including multiple sclerosis (MS), asthma and type1 diabetes. The 'hygiene hypothesis' postulates exposure to infectious agents confers protection against these disorders. One putative mechanism depends on the activity of regulatory T cells (Treg), naturally occurring or induced cells that prevent excessive immune activation and autoimmunity. Reports in the last 5 years lend credence to the hygiene hypothesis in MS: epidemiological investigations show an inverse relationship to infections with the nematode Trichuris, and a study with serial clinical, immunological and MRI follow-up shows MS patients developing intestinal parasitoses have much milder disease course compared with uninfected matched MS controls followed over 5 years. A role for Treg and also a novel population of B regulatory (Breg) cells is suggested in this study. The University of Nottingham has extensive experience with human parasite research and have completed essential safety studies of controlled infection with hookworm in normal volunteers and people with atopy. Asthma and Crohn's disease studies are underway and show an immunological effect even with 10 larvae. This is the first controlled parasite exposure study in patients with relapsing MS with in 36 patients 25 hookworm larvae vs 36 patients with placebo. Patients will be followed clinically (relapse rate, disability scores), immunologically and radiologically (serial MRI scans with Gadolinium) for 1 year. The cumulative number of new and active lesions on T2 weighted MRI will be the primary outcome measure. Regulatory network induction (Treg induction, Breg/Tr1 and NK) will be the immunological secondary outcome measure. Relapse rate will be secondary clinical outcome measure. A number of clinical, MRI and immune parameters will be exploratory measures. Cytokine profiles, eosinophil and egg counts, IgE and IgG subsets and IgE/IgG4 ratios will be measured, to relate altered immune responses to disease modulation. Immune responses will be assessed to neuroantigen and to mitogen, and parasite antigens (excretory/secretory products). This study will be an essential early step in assessing the potential for therapeutic immunomodulation with parasites in MS.

ELIGIBILITY:
Inclusion Criteria:

* Relapsing remitting MS (RRMS) (McDonald criteria) and secondary MS with super imposing relapse on condition that they fulfil the next conditions, MRI scan consistent with MS by Barkhof or Fazekas criteria
* Patients with at least 1 relapse in the last 12 months or 2 in the last 24 months;
* Patients with Expanded disability status scale (EDSS) score in the range of 0 to 5.5 at the screening and week 0 visit
* Patients of both genders, age >18 years and < 65 years
* Women of child bearing potential, (who have a negative pregnancy test) must agree to use methods of medically acceptable forms of contraception during the study.
* Be able and willing to comply with study visits and procedures per protocol.
* Understand and sign consent form at the screening

Exclusion Criteria:

No populations at risk of severe illness or death will be included in this study

* Life expectancy < 6 months.
* Patient is < 5 years free of malignancy, except treated basal cell skin cancer or cervical carcinoma in situ.
* Patient with grade III/IV cardiac problems as defined by the New York Heart Association Criteria. (i.e., congestive heart failure, myocardial infarction within 6 months of study)
* Patients with severe and/or uncontrolled medical condition.
* Pregnancy, lactation or intention to become pregnant during the course of the study (please also see above under inclusion criterion 5)
* Patient has a known diagnosis of human immunodeficiency virus (HIV) infection.
* Anaemia (Hb <10 g/dL for females, <11 g/dL for males)
* Prior or present evidence of parasitic infection; prior treatment with anti-helminthic drugs in the last 6 years.
* Patient with serious medical or psychiatric illness that could potentially interfere with the completion of the study treatment according to this protocol
* History of poor compliance or history of drug/alcohol abuse, or excessive alcohol consumption that would interfere with the ability to comply with the study protocol,
* Severe asthma, allergy, other autoimmune disease or any condition that the physician judges could be detrimental to subjects participating in this study; including deviations deemed clinically important from normal clinical laboratory

Previous treatment

* Treatment with interferon or glatiramer acetate within 8 weeks prior to baseline or immunosuppressive drugs within 12 weeks prior to baseline
* Treatment with bone marrow transplantation, total lymphoid irradiation, monoclonal antibodies (other than natalizumab, umbilical cord stem cells, AIMSPRO at any time prior to baseline
* Treatment with corticosteroids or ACTH within 4 weeks prior to baseline
* Treatment with any investigational agent within 12 weeks prior to baseline

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-12; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
The cumulative number of new or enlarging Gd+ lesions at month 9 | Month 9

SECONDARY OUTCOMES:
Percentage of cells positive simultaneously for CD4, CD25, foxp3 | End of trial
Cumulative number of newly active lesions (new GD+ T1; new and enlarging T2) at month 9 | Month 9
Change in expanded disability status scale (EDSS) at month 9 | Month 9

CONTACTS AND LOCATIONS:
Overall Officials: Cris Constantinescu, MD phD, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tanasescu R, Tench CR, Constantinescu CS, Telford G, Singh S, Frakich N, Onion D, Auer DP, Gran B, Evangelou N, Falah Y, Ranshaw C, Cantacessi C, Jenkins TP, Pritchard DI. Hookworm Treatment for Relapsing Multiple Sclerosis: A Randomized Double-Blinded Placebo-Controlled Trial. JAMA Neurol. 2020 Sep 1;77(9):1089-1098. doi: 10.1001/jamaneurol.2020.1118. PMID 32539079